CLINICAL TRIAL: NCT05735444
Title: Screening, Diagnosis and Treatment of Obstructive Sleep Apnea Syndrome in Hypertensive Patients in China: A Prospective National Multi-center Registry
Brief Title: Prospective National Multi-center Registry of Obstructive Sleep Apnea Syndrome in Hypertensive Patients in China
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension and the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Other Study IDs: OSA-HT
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: Hypertension; Obstructive sleep apnea syndrome; Continuous positive airway pressure; Registry
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — We collect 20 ml of venous blood and 20 ml of urine at baseline and the end of follow-up, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure (CPAP) is one of the standard medical treatments for patients with OSAS. The mechanism of CPAP probably involves maintenance of a positive pharyngeal transmural pressure so that the intraluminal pressure exceeds the surrounding pressure. CPAP also increases end-expiratory lung volume, which stabilises the upper airway through caudal traction.

SUMMARY:
Study name: Screening, Diagnosis and Treatment of Obstructive Sleep Apnea Syndrome in Hypertensive Patients in China: A Prospective National Multi-center Registry.

Rationale: Obstructive sleep apnoea syndrome (OSAS) is a common secondary cause of hypertension and significantly correlated with the risk of cardiovascular and cerebrovascular diseases. However, continuous positive airway pressure (CPAP) only shows modest blood pressure lowering effect, although it is effective in the relieve of daytime sleepiness and other symptoms of OSAS. One of the possible reasons for the low antihypertensive efficacy might be the low adherence to CPAP therapy. Nonetheless, few studies systematically investigated CPAP adherence with regard to its prediction and clinical relevance for cardiovascular protection and prevention.

Objective: 1) To evaluate short- and long-term CPAP adherence in patients with hypertension and obstructive sleep apnea syndrome; 2) To investigate the predictors of short- and long-term CPAP adherence; 3) To explore the correlation between the CPAP adherence and blood pressure, target organ damage and the incidence of cardiovascular and cerebrovascular events.

Study design: Prospective, multi-center, observational study.

Study population: Patients with hypertension who are suspected to have obstructive sleep apnea syndrome due to snoring, daytime sleepiness and other related symptoms are considered eligible and should meet the following criterias: 1) Agree to participate in the study and sign the informed consent; 2) At least 18 years old; 3) STOP-Bang questionnaire, score ≥3 points; 4) Complete polysomnography in hospital; 5) Currently on CPAP therapy.

Follow up: 3, 6 and 12 months after registry.

Sample size estimation: At least 633 patients.

Timeline: Start of subjects' enrollment: Jan 2023; End of subjects' enrollment: December 2026; End of study: December 2026.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
Study name: Screening, Diagnosis and Treatment of Obstructive Sleep Apnea Syndrome in Hypertensive Patients in China: A Prospective National Multi-center Registry.

Rationale: Obstructive sleep apnoea syndrome (OSAS) is a common secondary cause of hypertension and significantly correlated with the risk of cardiovascular and cerebrovascular diseases. However, continuous positive airway pressure (CPAP) only shows modest blood pressure lowering effect, although it is effective in the relieve of daytime sleepiness and other symptoms of OSAS. One of the possible reasons for the low antihypertensive efficacy might be the low adherence to CPAP therapy. Nonetheless, few studies systematically investigated CPAP adherence with regard to its prediction and clinical relevance for cardiovascular protection and prevention.

Objective: 1) To evaluate short- and long-term CPAP adherence in patients with hypertension and obstructive sleep apnea syndrome; 2) To investigate the predictors of short- and long-term CPAP adherence; 3) To explore the correlation between the CPAP adherence and blood pressure, target organ damage and the incidence of cardiovascular and cerebrovascular events.

Study design: Prospective, multi-center, observational study.

Study population: Patients with hypertension who are suspected to have obstructive sleep apnea syndrome due to snoring, daytime sleepiness and other related symptoms are considered eligible and should meet the following criterias: 1) Agree to participate in the study and sign the informed consent; 2) At least 18 years old; 3) STOP-Bang questionnaire, score ≥3 points; 4) Complete polysomnography in hospital; 5) Currently on CPAP therapy.

Follow up: 3, 6 and 12 months after registry.

Sample size estimation: At least 633 patients.

Timeline: Start of subjects' enrollment: Jan 2023; End of subjects' enrollment: December 2026; End of study: December 2026.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in the study and sign the informed consent;
2. At least 18 years old;
3. STOP-Bang questionnaire, score ≥3 points;
4. Complete polysomnography in hospital;
5. Currently on CPAP therapy.

Exclusion Criteria:

1. Clinic systolic/diastolic blood pressure ≥180/110 mmHg;
2. Previous or current treatment for OSAS without CPAP;
3. Severe respiratory diseases such as chronic obstructive pulmonary disease, or contraindications to CPAP therapy, such as pneumothorax, pulmonary bulla and new-onset stroke；
4. Sleep disorders or insomnia;
5. Intolerance of CPAP therapy;
6. Patient with cognitive dysfunction who are unable to provide informed consent;
7. Other circumstances that patients are not appropriate for the study upon the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension who are suspected to have obstructive sleep apnea syndrome due to snoring, daytime sleepiness and other related symptoms are considered eligible and should meet all the inclusion criterias but not any of the exclusion criterias.
Sampling Method: Non-Probability Sample
Enrollment: 633 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean 24-hour ambulatory blood pressure after 12-month CPAP treatment from baseline | 12 months
  Units on a mm Hg

SECONDARY OUTCOMES:
Change in mean daytime ambulatory blood pressure after 12-month CPAP treatment from baseline | 12 months
  Units on a mm Hg
Change in mean nighttime ambulatory blood pressure after 12-month CPAP treatment from baseline | 12 months
  Units on a mm Hg
Change in mean clinic blood pressure after 12-month CPAP treatment from baseline | 12 months
  Units on a mm Hg
Change in mean home blood pressure after 12-month CPAP treatment from baseline | 12 months
  Units on a mm Hg
Change in brachial-ankle pulse wave velocity after 12-month CPAP treatment from baseline | 12 months
  Units on a cm/s
Change in left ventricular mass index after 12-month CPAP treatment from baseline | 12 months
  Unit on a g/m^2
Change in urine albumin-creatinine ratio after 12-month CPAP treatment from baseline | 12 months
  Unit on a mg/mmol

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided